CLINICAL TRIAL: NCT06930781
Title: Evaluation of Clinical Outcomes of Ponto Procedures Performed in Settings Outside the Main Operating Room (i.e. Out-of-OR)
Status: Recruiting | Type: Observational
Sponsor: Oticon Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: BC118; CIV-ID 25-01-051014 (Other: Swedish Medical Products Agency)
Record Dates: First submitted 2025-04-01; First posted 2025-04-16 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Hearing Loss; Bone Anchored Hearing Aids
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Retrospective group: Data gathered from retrospective chart reviews of patients who have undergone Ponto-implantation in an out-of-OR setting from 2019 and onwards
  Interventions: Device: Ponto implantation
- Prospective group: Patients who have undergone Ponto implantation in an out-of-OR setting and participated in the study by filling out questionnaires.
  Interventions: Device: Ponto implantation

INTERVENTIONS:
Device: Ponto implantation — Ponto implantation is a surgical procedure to implant a bone-anchored hearing device, improving hearing by transmitting sound directly to the inner ear through bone conduction.

SUMMARY:
This study is a combined retro- and prospective, single arm, multicentre investigation designed to follow clinical practice for Ponto-implantations performed out of OR. The overall objective is to investigate the complication rate for procedures performed out-of-OR.

DETAILED DESCRIPTION:
The study is observational and non interventional and follows clinical practice at participating clinics with the only exception of three questionnaires given to consenting patients after surgery and during follow-up, after loading of the sound processor.

The study is a combined retro- and prospective study. The retrospective part consists of a chart review of patients who have undergone Ponto-implantation out of OR from 2019 and onwards. The prospectively recruited subjects are patients who are planned to undergo Ponto-implantation surgery out-of-OR.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥18 years old) undergoing Ponto implantation in an out-of-OR setting from 2019 and onwards
* Signed informed consent (applicable for subjects answering questionnaires)

Exclusion Criteria:

* No exclusion criteria have been set for this observational investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Bone-conduction hearing device users
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-05-07 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative complications at surgery | During the Ponto-implantation surgery

SECONDARY OUTCOMES:
Assessment of procedure room variables | 12 months after study start
  To make an assessment of how procedure rooms that are used for Ponto out-of-OR surgeries look like. Will be measured using the 'Procedure room used for Out-of-OR Ponto-surgery questionnaire'
To assess surgical parameters | During Ponto-implantation surgery
  With this outcome, the aim is to assess the surgical variables present during Ponto out-of-OR surgeries. A series of yes or no questions will be presented in a form to the surgeon regarding the use of anesthesia, sedatives, implants, and abutments of different lengths. The results will be presented in a table.
Evaluation of patient experience of surgical procedure based on Ponto procedure questionnaire | 5-10 days after Ponto surgery
  Score is reported on a scale of 5 steps, were the lowest value (1) is the worst and the highest value is the best (5)
To assess postoperative events and complications | From day of surgery, through study completion, an average of 1 year
  All postoperative events and complications will be presented in a descriptive table, listing how many were affected by each type of event or complication.
To assess rate of implant survival | 3 months after surgery, and through study completion, an average of 1 year.
  Implant survival will be assessed at least once, at 3 months. If follow-up data is available, implant survival will be assessed through study completion, an average of 1 year.
To assess time from surgery to sound processor loading | Time from surgery to sound processor loading which happens at an average of 3 months after surgery.
To assess sound processor usage time | 3 months after surgery, and through study completion, an average of 1 year.
To assess effectiveness of hearing rehabilitation using IOI-HA questionnaire | 3 months after surgery
  Will be assessed using the standardised questionnaire International Outcome Inventory for Hearing Aids (IOI-HA) score at 3 months post-surgery. In the questionnaire, each item has five response choices proceeding from the worst outcome to the best outcome (1-5). The score will be presented as mean score with, standard deviation and median for the two groups.
To assess patient-reported benefit after BAHS treatment using the questionnaire Glasgow Benefit Inventory (GBI) | 3 months after surgery
  Glasgow Benefit Inventory (GBI) benefit scores will be presented for total-, general-, social- and physical scores at 3 months post-surgery. The GBI uses a scale from -100 to +100, where scores above 0 indicate improved quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Dr David Morris, Principal Investigator — Queen Elizabeth II Health Sciences Centre
Locations (2):
- Sweden (2):
  - Sunderby Sjukhus, Luleå, Norrbotten County
  - Skåne University Hospital, Lund, Skåne County